CLINICAL TRIAL: NCT01089829
Title: The Pathological Relationships Between Chronic Kidney Disease (CKD)and the Development of Lower Limb Threatening Complications
Brief Title: Risk Factors for Foot Ulceration in the Chronic Kidney Disease (CKD) Population
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cardiff University (Other)
Collaborators: Podiatry Department, Cardiff & Vale University Health Board (Unknown); School of Health Sciences, UWIC (Unknown); Institute of Nephrology, Cardiff & Vale University Health Board (Unknown)
Responsible Party: Dr Stephen Riley, Senior Lecturer and Hon Consultant Nephrologist
Other Study IDs: SRiley&NJones
Record Dates: First submitted 2010-02-04; First posted 2010-03-19 (Estimated); Last update posted 2010-03-19 (Estimated); Status verified 2010-01

CONDITIONS: Chronic Kidney Disease
Keywords: CKD; Foot Ulceration; Diabetes
MeSH Terms: conditions — Renal Insufficiency, Chronic; Foot Ulcer; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CKD Stage 4: eGFR <30
  Interventions: Other: Foot examination
- CKD Stage 5: Receiving Haemodialysis or Peritoneal dialysis therapy
  Interventions: Other: Foot examination

INTERVENTIONS:
Other: Foot examination — Non-invasive neurological sensory testing
  Non-invasive doppler assessment of peripheral arterial system
  Other Names: CKD Stage 4 interventions at baseline, 12 & 24 months; CKD Stage 5 interventions at baseline, 6 & 12 months

SUMMARY:
Foot ulceration is a risk factor that has been associated with early death in patients with chronic kidney disease. Little is known about the relationship between these risk factors that develop in patients with kidney failure and the onset of lower limb threatening foot ulcers.

Diabetes is a major cause of both kidney disease and foot ulceration; however a previous study reported that a significant proportion of kidney failure patients on haemodialysis treatment without a diagnosis of diabetes also had these risk factors that could lead to foot ulceration.

The aim of this study will be to identify these risk factors associated with lower limb threatening disease in patients with advanced kidney failure. In addition a robust screening tool will be developed to address the reliability and validity of current screening methods deemed to be gold standard in the assessment of diabetic foot disease in this Chronic Kidney Disease population.

It is important to follow the progression of these risk factors as the kidney failure worsens. The study also intends to screen patients as they start dialysis treatment and follow their progress with respect to risk factors known to predispose to foot ulceration over their first year of treatment. The proposed outcome from this study is to develop a strategy to identify patients with kidney failure that are at risk of foot ulceration and intervene at an early point to prevent the life threatening complications associated foot disease.

DETAILED DESCRIPTION:
The risk factors contributing to foot ulceration in the diabetic population are well published, and an abundance of these publications demonstrate the acceleration of risk factors in association with diabetic nephropathy.

It is also apparent that there are risk factors present in the non-diabetic Chronic Kidney Disease population but much less information about there prevalence and progression is published. A recent pilot study reported significant risk factors for foot ulceration in a population of subjects receiving haemodialysis therapy in the absence of diabetes mellitus.

The study will aim to increase the understanding of Chronic Kidney Disease (CKD) and the development of foot ulceration in the diabetic and non-diabetic Chronic Kidney Disease population as renal failure progresses and dialysis is initiated.

Design and methodology:

Patient Identification:

It is proposed to identify patients with Chronic Kidney Disease level 4 (renal function at between 15 and 30% of normal)in the Nephrology clinics at University Hospital of Wales, Cardiff. It is this group of patients that are most at risk of progression of renal disease towards end stage and subsequent need for dialysis.

A proportion of the patients will be identified from the pre-dialysis clinics that are due to commence dialysis imminently. It is this group of patients that will used to examine the specific effects of dialysis modality on risk factors for foot ulceration The directorate of Nephrology and Transplantation in Cardiff has 450 haemodialysis patients, 140 peritoneal dialysis (CAPD) patients, and around 400 Chronic Kidney Disease level 4 patients. Approximately 100 new patients commence dialysis each year of which 35 will start peritoneal dialysis and the rest haemodialysis.

Renal patients currently have the freedom to choose their preferred modality of dialysis following a series of informed consultations with the Physician. One method may be indicated over another if the patient does not meet the suitability criteria for one or other of the modalities. However, current recruitment trends demonstrate that most patients prefer to choose haemodialysis despite the socioeconomic challenges the therapy poses on their quality of life and the cost constraints on the health service.

A previous study demonstrated that 20% of patients with diabetes develop foot ulceration within the first year of commencing haemodialysis and this may be attributed to the hypoxia of the peripheral tissues during the haemodialysis process. There is much less information about the changes seen with the initiation of peritoneal dialysis and this study may help to influence dialysis modality choice in the future if one method of dialysis is associated with the development of fewer lower limb threatening complications.

Inclusion criteria: Stage 4/5 Chronic Kidney Disease (eGFR <30ml/min) Over 18 years of age Exclusion criteria: Chronic Kidney Disease Stage 1-3 (eGFR >31) Inability or refusal to give informed consent Life expectancy < 6 months

The Proton database held within Nephrology along with clinic lists will be used to identify potential patients by the research team and an invitation letter will be sent with a study information leaflet prior to their clinic visit.

The Physician in the clinic will recruit the patient to take part in the study during the Outpatient consultation. Clinic lists will also be reviewed to identify patients with Chronic Kidney Disease stage 4/5.

Screening protocol:

The longitudinal prospective study proposed would expand on pilot study results to include level 4 Chronic Kidney Disease and monitor the development of lower limb threatening risk factors with the progression of kidney failure towards end stage renal disease.Patients will be followed for a 2 year period.

A single Podiatrist will undertake the interview and use non-invasive techniques to assess feet for physiological risk factors in accordance with evidence-based practice.

The Renal Foot Screening Tool has been developed and will be used to prospectively identify the neurovascular risk factors for foot ulceration.

Patients would have podiatry assessment at baseline, 12 and 24 months. In addition a triggered assessment would take place at commencement of dialysis.

Power calculations are difficult to undertake given the lack of current knowledge of risk factors for this group of patients. Following consultation with a statistician on the supervisory team the minimum figure of 100 has been adopted as the target for Chronic Kidney Disease level 4 patients with an additional minimum 100 patients commencing renal replacement therapy over the course of the study period.The target for recruitment was estimated taking into account the financial and resource implications, and was agreed by the supervisory team to be a realistic sample size. Subsequent statistical analysis will include multiple regression.

Interview:

Demographic and medical information will be obtained through patient interview and medical records at the time of the foot screening.

Patients will be questioned about prior foot care education, patient perception of their current foot health status, history of Podiatry care, history of foot ulceration and previous amputation.

Non-invasive assessment techniques

No current foot screening provision for patients with Chronic Kidney Disease exists in Cardiff.

The research participants will have a detailed foot screening consultation that will identify potential risks of foot ulceration allowing earlier intervention should it be required.

The patients enrolled into this study will have enhanced care in terms of identification of potential foot ulceration. However, this does raise some ethical concerns. The first is that patients may be seen at presentation with a foot ulcer or be at high risk of developing a foot ulcer and these patients will be referred to the Podiatry service for routine treatment. The other issue is that patients will not be given verbal education regarding their specific foot care needs during the contacts. We justify this in that we are trying to find the factors associated with Chronic Kidney Disease that contribute to foot ulceration in a longitudinal fashion. Intervention with education could confound the true prevalence for the study. We would acknowledge that simply checking the feet of a patient would alter their awareness and this also may influence the study findings in a small way. Information leaflet provided to each high risk participant will give indications of the danger signs that can preceded to ulceration and infection,with a help line telephone number to call should a participant develop any of these warning signs.

The participant will be fast track referred to the Cardiff & Vale Podiatry department, and given an urgent appointment at a Cardiff & Vale Podiatry Wound Clinic for a treatment plan. Follow up care will be provided by the local Community Podiatry Service after the wound has healed.

Non-healing foot ulcers will be referred to the Multi-disciplinary Foot Ulcer Clinic for review by the Vascular, Orthopaedic, and Medical team.

Peripheral neuropathy:

To ensure all patients with neuropathy are identified multiple forms of assessment will be used for each patient. All methods of assessment are standardised, and any tests will be demonstrated on the back of one hand for the patient to experience prior to formal neuropathy testing.

The previously published Neuropathy Symptom Score is used to pick up symptomatic peripheral neuropathy. This scoring system is used to identify the sensory symptoms of peripheral neuropathy, such as aching, burning, prickling, numbness, and sharp pain.

Light pressure sensation is tested using the Semmes-Weinstein 10g monofilament at 10 sites on each foot. The patient is instructed to close their eyes, the 10g monofilament is applied at a 90 degree right angle to the selected site until it buckled, and held for 1 second before moving onto the next test site.

A positive neuropathy score for the monofilament assessment is defined as inability to perceive the monofilament sensation on the testing sites on each foot.

A neurothesiometer is used to test vibration perception threshold. This device is applied with the tractor balanced vertically onto the pulp of the hallux with the voltage increased at the base unit until the patient can perceive the vibration sensation. A mean of three readings would be recorded for each foot.A value of 25 volts and over would confirm the patient being 'At Risk' of foot ulceration.

Given that patients often score differently for each test, patients with a positive score during any of the 3 repetitions are classified as having peripheral neuropathy.

Vascular Insufficiency:

The Edinburgh Claudication Questionnaire is used to diagnose symptomatic vascular insufficiency. Patients score positive for symptomatic vascular insufficiency if they described either symptoms of intermittent claudication or rest pain. The possibility of concomitant peripheral neuropathy in this patient population is such that symptoms alone are insufficient to diagnose peripheral vascular disease. Therefore a hand held Doppler ultrasound is used to locate the dorsalis pedis and posterior tibial arteries. The probe is lightly applied to the skin to avoid occlusion of the artery, and the audible sound is reproduced on a printout in preparation for waveform analysis.

Arterial insufficiency is recorded when both the dorsalis pedis and posterior tibial signals are monophasic in a single lower limb.

Foot Pathology:

It is recognised that foot pathology is an additional risk factor for foot ulceration especially in those patients with either peripheral neuropathy or vascular insufficiency.

Both feet are visually inspected for common pathologies predisposing to diabetic foot ulceration. Any deformity, including hammer toes and Charcot deformity, nail dystrophies, corns and calluses are reported as additional risk factors.

The presence of active foot ulceration is documented and graded according to the Texas Wound Classification system to ascertain the severity of the wounds presenting within a cohort.

Data collected on laptop will only have study identification number recorded to ensure the anonymisation of participants during data collection and data analysis by the research team statistician. The laptop will be password secure and be stored in a locked filling cabinet in a locked office with key access to the Band 7 Podiatrist. Files containing consent forms will be indexed in numerical order of study identification numbers, and will be stored in a locked filling cabinet with only access to the Principle Investigator and the Band 7 Podiatrist. The file will be the only source of person identifiable information.

Body Composition Monitoring:

The use of a none invasive assessment of body composition will allow a review of body fluid status which may impact on the ability of tissues to heal.

Resources:

A Podiatrist will be required to undertake this longitudinal study on a part time basis. This is supported by the fact that the highly specialised skills developed by the Podiatrist need to be maintained during the PhD study period also require a contribution of specialist clinical duties.

The equipment needed to make the measurements is available from the department of Podiatry and is calibrated and used on a day to day basis for current patient care.

Willing participants will be offered foot screening at the end of the Nephrology OPD consultation to minimise any further inconvenience with travelling and parking costs A contribution may be required for patients travelling expenses when they are recalled.

The full support of the Institute of Nephrology has been obtained in terms of supervision by a Consultant Nephrologist and access to patient information.

Dissemination:

It is proposed that this work will be presented at Podiatry and Renal conferences in the UK and overseas. Minimum of 3 papers and 3 conference presentations. There is room for publication in Podiatry and Renal publications to ensure both groups of professionals are informed. Posters will be prepared for international conferences. There is also an opportunity to consider Nursing conferences to raise general awareness of the issue, and any opportunities that arise for the preparation of review articles will be taken.

Outcomes and impact:

The primary outcome of the study is to identify the neurovascular risk factors for foot ulceration as renal function declines, and to develop a suitable foot protection programme for Chronic Kidney Disease patients. The secondary outcome measure is to identify whether dialysis modality choice influence foot ulcer development and should this be used to inform patient choice of dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Stage 4/5 Chronic Kidney Disease (EGFR <30ml/min) Over 18 years of age

Exclusion Criteria:

* CKD stage 1-3 (eGFR >31)
* Inability or refusal to give informed consent
* Life expectancy < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is proposed to identify patients with CKD level 4 (renal function at between 15 and 30% of normal)in the Nephrology clinics at University Hospital of Wales, Cardiff. It is this group of patients that are most at risk of progression of renal disease towards end stage and subsequent need for dialysis.
  A proportion of the patients will be identified from the pre-dialysis clinics that are due to commence dialysis imminently. It is this group of patients that will used to examine the specific effects of dialysis modality on risk factors for foot ulceration The directorate of Nephrology and Transplantation in Cardiff has 450 haemodialysis patients, 140 peritoneal dialysis (CAPD) patients, and around 400 CKD level 4 patients. Approximately 100 new patients commence dialysis each year of which 35 will start CAPD and the rest haemodialysis.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-04; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of the study is to identify the neurovascular risk factors for foot ulceration as renal function declines, and to develop a suitable foot protection programme for CKD patients. | 4 years

SECONDARY OUTCOMES:
The secondary outcome measure is to identify whether dialysis modality choice influence foot ulcer development and should this be used to inform patient choice of dialysis. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Ian DR Mathieson, Study Director — School of Health Sciences, UWIC
Locations (1):
- University Hospital of Wales, Cardiff, United Kingdom, United Kingdom